212458 (MENACWY=ccl -001 PRI) Statistical Analysis Plan Amendment 5

| , | Statistical Analysis Plan |
|---|---|
| Title: | A Phase I/II, randomised, controlled study to assess<br>the safety, effectiveness and immune response of<br>meningococcal combined ABCWY vaccine when<br>administered to healthy adults (Phase I) and to healthy<br>adolescents and adults (Phase II). |
| eTrack study number and<br>Abbreviated Title | 212458 (MENACWY=cci -001 PRI) |
| Scope: | All analyses for the primary and secondary objectives of the study and interim analysis. The analysis details for tertiary objectives are described in separate Statistical Analysis Plan (SAP). |
| Date of Statistical Analysis<br>Plan | Amendment 5 Final: 29 Aug 2023 |

APP 9000058193 Statistical Analysis Plan Template V5 (Effective date: 1July2020)

212458 (MENACWY=ccl -001 PRI) Statistical Analysis Plan Amendment 5

### **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | T OF A | BBREVIATIONS | | 7 |
| 1. | DOCU | MENT HISTORY | | 8 |
| 2. | OBJE | CTIVES/ENDPOINTS | | 10 |
| 3. | STUD | V DESIGN | | 16 |
| ٥. | 3.1. | | | |
| | 0 | | design | |
| | | 3.1.2. Phase II study | design | 18 |
| | | 3.1.2.1. Ph | ase II: Formulation and Schedule-finding | 18 |
| | | 3.1.2.2. Ph | ase II: Sourcing | 20 |
| 4. | ANAL | YSIS SETS | | 23 |
| | | | | 21 |
| 5. | STAT | STICAL ANALYSES | | 28 |
| | 5.1. | | | |
| | | | sposition of subjects | |
| | 5.2. | | and baseline characteristics | |
| | | | ned in the protocol | |
| | 5.3. | | siderations | |
| | 5.5. | CCI | | 29 |
| | | | | 29 |
| | | | | 29 |
| | | | | 30 |
| | | | | 30 |
| | | | | 30 |
| | | | | 31 |
| | | | | 32 |
| | | 5.3.2. Additional con | siderations | |
| | | CCI | old of dillotte | |
| | 5.4. | Secondary endpoints | | |
| | | | ned in the protocol | |
| | | 5411 Ph | ase L (Safety Lead-in) | 34 |
| | | CCI | | 35 |
| | | | | 35 |
| | | | | 33 |
| | | | | 35 |

| | | | ı | | :12458 (MENACWY= <mark>cci</mark><br>Statistical Analysis Plan <i>I</i> | |
|---|---|---|---|---|---|---|
| | | | | | | 26 |
| | | | 5.4.1.3. | Phase II (Sourcing) | | 36<br>36 |
| | 5.5. | CCI | J. <del>4</del> . 1.J. | Thase if toourcing | | 37 |
| | 5.5. | | | | | 37 |
| | | | | | | 37 |
| | | | | | | 37 |
| | | | | | | 37 |
| | | | | | | 37 |
| | | | | | | 38 |
| | | | | | | 38 |
| | | | | | | 38 |
| | | | | | | 30 |
| | | | | | | 38 |
| | CCI | | | | | |
| 6. | | | | | | 39 |
| 7. | | | | | | 40 |
| | | | | | | 40 |
| | | | | | | 41 |
| _ | | | | | | 4.4 |
| 8. | | | | | | 41 |
| 9. | | | | | | |
| 9. | | | | | | 41 |
| | 9.1. | Data de | rivation | | | |
| | 9.1. | | | | | |
| | J.Z. | 9.2.1. | | | | |
| | | 9.2.2. | | | | |
| | | 0.2.2. | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | _ |
| 10. | ANNE | XES | | | | 42 |
| | CCI | | | | | 42 |
| | | | | | | 42 |
| | | | | | | 42 |
| | | | | | | 42 |
| | | | 10.1.2.3. | | icited events | |
| | | | 40.45.4 | | with electronic diaries | |
| | | 40.4.0 | 10.1.2.4. | | events | |
| | | 10.1.3. | | | | |
| | | | 10.1.3.1. | | ays | |
| | | | 10.1.3.2.<br>10.1.3.3. | | onthsears | |
| | | | 10.1.3.3. | Aye at 111 St 40SE 111 YE | aı 5 | 44 |

| | CONFIDENTIAL 212458 (MENACWY=column)-0 | |
|--------------------|-------------------------------------------------|----|
| | Statistical Analysis Plan Amen | |
| | Weight | |
| | Height | |
| | Body mass index (BMI) | |
| | Temperature | |
| 10.1.3.8. | Numerical serology results | 45 |
| 10.1.3.9. | ( ) | |
| | concentrations (GMCs) | |
| | Calculation of the 4-fold rise | |
| | Onset day | |
| | Duration of events | 46 |
| 10.1.3.13. | Counting rules for combining solicited and | |
| | unsolicited adverse events | 46 |
| 10.1.3.14. | Counting rules for occurrences of solicited | |
| | events | |
| 10.1.4. Display of | decimals | 46 |
| 10.1.4.1. | Percentages | 46 |
| | Differences in percentages | |
| | Demographic/baseline characteristics statistics | |
| | Serological summary statistics | 48 |
| CCI | | 48 |
| | | 48 |
| | | 48 |
| 11. REFERENCES | | 48 |

212458 (MENACWY=ccl -001 PRI) Statistical Analysis Plan Amendment 5

### **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study groups, intervention and blinding – Phase I | 18 |
| Table 2 | Study groups, intervention and blinding – Phase II (Formulation and Schedule-finding) | 20 |
| Table 3 | Study groups, intervention and blinding – Phase II (Sourcing) | 22 |
| Table 4 | Analysis sets | 23 |

212458 (MENACWY=ccl -001 PRI) Statistical Analysis Plan Amendment 5

### **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1 | Study design overview – Phase I (Safety Lead-in) | 17 |
| Figure 2 | Study design overview – Phase II (Formulation and Schedule-finding) | 19 |
| Figure 3 | Study design overview – Phase II (Sourcing) | 21 |
| Figure 4 | Hierarchical testing of hypothesis | 39 |

212458 (MENACWY=ccl -001 PRI) Statistical Analysis Plan Amendment 5

#### LIST OF ABBREVIATIONS

**AE** Adverse event

**AESI** Adverse Events of Special Interest

ANCOVA Analysis of Covariance
ANOVA Analysis of Variance
CI Confidence Interval

**CRF** Case Report Form

CTRS Clinical Trial Registry Summary

EL.U/mL ELISA unit per millilitre

Eli Type Internal database code for type of elimination code

**ELISA** Enzyme-linked immunosorbent assay

**ES** Exposed Set

**FAS** Full Analysis Set

**F&SF** Formulation and Schedule-finding

**GMC** Geometric mean antibody concentration

**GMT** Geometric mean antibody titre

**GSK** GlaxoSmithKline

**HR** Hazard Ratio

IU/mL International units per millilitre

LL Lower Limit

**MedDRA** Medical Dictionary for Regulatory Activities

NA Not Applicable

**PDMP** Protocol Deviation Management Plan

PPS Per-Protocol Set

**RR** Relative Risk

SAE Serious adverse event
SAP Statistical Analysis Plan

SBIR GSK Biologicals Internet Randomisation System

**SD** Standard Deviation

**SDTM** Study Data Tabulation Model

SR Study Report

SUSAR Suspected Unexpected Serious Adverse Reaction

UL Upper Limit

### 1. DOCUMENT HISTORY

| Date | Description | Protocol<br>Version |
|---|---|---|
| 02 June 2021 | First Version | Final: 15<br>January 2021 |
| 22 July 2021 | <ul> <li>Tdap has been replaced with placebo in the phase II formulation and schedule finding</li> <li>Update of the number of participants enrolled in the phase II formulation and schedule finding (change of testing strategy, split of the alpha, cf. to the protocol for more details)</li> <li>Update of number of participants enrolled in the phase II Sourcing and the age range for inclusion criteria</li> </ul> | Amendment 2:<br>24 June 2021 |
| 19 October<br>2021 | <ul> <li>In the Phase II Formulation and Schedule finding, the participants in the Control group will have no study intervention at Visit V3 (Month 4). This visit (Visit V3) has been replaced by a phone call (TC).</li> </ul> | Amendment 3:<br>28 September<br>2021 |
| 11 May 2022 | <ul> <li>Amendment 3</li> <li>Two dosing schedules have been added in the Phase II Sourcing part, leading to changes in study design and to some objectives and endpoints</li> <li>Detailed definition populations by phases</li> </ul> | Amendment 4:<br>22 March 2022 |
| 06 June 2023 | <ul> <li>Minor corrections throughout the document to improve clarity</li> <li>Section 4.2: Exclusion criteria for FAS were made explicit</li> <li>Section 4.2: All the exclusion criteria for PPS were corrected (when needed) and split by phase of the study</li> <li>Section 5 – Statistical analyses: It was added a subsection 5.1 – Disposition of subjects. Therefore, the following subsections have been renumbered (e.g., 5.1 became 5.2, etc.)</li> </ul> | Amendment 4:<br>22 March 2022 |

| | Statistical Analysis | Plan Amendment 5 |
|---|---|---|
| | Section 5.2 (formerly 5.1): description of analyses for demography were corrected | |
| | Section 5.3 (formerly 5.2) – Primary analyses: categorization of each AESI either as a new onset condition or as an exacerbation of a pre-existing chronic condition (as proposed by CBER) is documented in each "Safety" subsection | |
| | Section 5.4 (formerly 5.3): removal of the sentence "The 95% CIs for the difference in percentages between ABCWY groups and control group will be constructed using the method of Miettinen and Nurminen", as the respective objective does not involve any difference. Column | |
| | • | |
| | Subsection 10.1.3: definitions of GMT and GMC were rephrased new subsection with updated 4-fold rise definition amendment of rules on how to address possible incoherence in e-diary-recorded solicited administration site adverse events | |
| | Subsection 10.1.4: rules for the display of decimals have been corrected / clarified | |
| 29 Aug 2023 | Amendment 5 | Amendment 4: |
| | Section 4.2: All the criteria for eliminating data from analysis sets have been reformulated using categories and subcategories of the PDMP, as per new process | 22 March 2022 |
| | Section 6: Figure 4 has been re-made to add one arrow that goes from the right column to the left column | |
| | Subsection 10.1.3.14: Counting rules to address ambiguities in e-diary-recorded solicited administration site adverse events have been better detailed | |

212458 (MENACWY=ccl -001 PRI) Statistical Analysis Plan Amendment 5

### 2. OBJECTIVES/ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Phase I – Safety lead | I-in, Dose escalation |
| Prir | nary |
| To evaluate the safety and reactogenicity of the 2 formulations (cc) vaccine. | The frequencies and percentages of participants with solicited administration site and systemic events during the 7 days (including the day of vaccination) following each vaccination at Day 1 and Day 31 in all groups. |
| | The frequencies and percentages of participants with any unsolicited AEs (including all SAEs, AEs leading to withdrawal, and AESIs) during the 30 days (including the day of vaccination) following each vaccination at Day 1 and Day 31 in all groups. |
| | <ul> <li>The frequencies and percentages of participants<br/>with SAEs, AEs leading to withdrawal and AESIs<br/>throughout the study period in all groups (Day 1<br/>through Day 211).</li> </ul> |
| | The frequencies and percentages of participants with haematological and biochemical laboratory abnormalities, and changes from the baseline values, after the first vaccination at Day 8, in all groups. |
| Phase II – Formulation | n and Schedule-finding |
| | nary |
| To demonstrate the superiority of the effectiveness of the vaccine (cc) ) when administered at 0,2- or 0,6-months schedule, compared to the MenB vaccine administered at 0,6-months schedule*. | The percentages of samples with bactericidal serum activity using enc-hSBA against a panel of 110 randomly selected endemic US <i>N. meningitidis</i> serogroup B invasive disease strains at 1 month after the last vaccination (Day 211, Month 7) in all groups. |
| To demonstrate the immunological non-inferiority of the vaccine (columns) administered at 0,2- or 0,6-months schedule compared to the MenACWY vaccine (single dose)*;†. | The percentages of participants achieving a 4-fold rise** in hSBA titres against serogroups A, C, W and Y at 1 month after the |
| raceine (emgie acce) | • last column vaccination (Day 211, Month 7) for the ABCWY groups and, |
| | MenACWY vaccination (Day 31, Month 1) in the Control group, relative to Day 1, Month 0 in CO |
| | and Control groups and relative to 3 months pre-first column vaccination (Day 31, Month 1) in column groups. |

| Objectives | Endpoints |
|---|---|
| To evaluate the safety and reactogenicity of the vaccine (science), the MenB vaccine and the MenACWY vaccine. | <ul> <li>The frequencies and percentages of participants<br/>with solicited administration site and systemic<br/>events during the 7 days (including the day of<br/>vaccination) following each vaccination at:</li> </ul> |
| | Day 1, Day 121 and Day 181 in the groups, and |
| | Day 1 and Day 181 in the Control group |
| | The frequencies and percentages of participants with any unsolicited AEs (including all SAEs, AEs leading to withdrawal, and AESIs) during the 30 days (including the day of vaccination) following each vaccination at: |
| | <ul> <li>Day 1, Day 121 and Day 181 in the</li> <li>groups,</li> <li>and</li> </ul> |
| | <ul> <li>Day 1 and Day 181 in the Control group.</li> </ul> |
| | <ul> <li>The frequencies and percentages of participants<br/>with SAEs, AEs leading to withdrawal and AESIs<br/>throughout the study period in all groups (Day 1<br/>through Day 541).</li> </ul> |
| | -Sourcing |
| | nary |
| To evaluate the safety and reactogenicity of the 2 formulations (CCI vaccine.) of the CCI vaccine. | The frequencies and percentages of participants with solicited administration site and systemic events during the 7 days (including the day of vaccination) following each vaccination at: |
| | <ul> <li>at Day 1 and Day 31 in groups,</li> </ul> |
| | – at Day 1 and Day 61 in <b>ccl</b><br>groups, and |
| | – at Day 1 and Day 181 in <mark>ccl</mark><br>groups. |
| | The frequencies and percentages of participants with any unsolicited AEs (including all SAEs, AEs leading to withdrawal, and AESIs) during the 30 days (including the day of vaccination) following each vaccination at: |
| | <ul><li>at Day 1 and Day 31 ccl<br/>groups,</li></ul> |
| | – at Day 1 and Day 61 in <b>cel</b><br>groups, and |
| | – at Day 1 and Day 181 in <mark>ccl</mark><br>groups. |

| | Statistical Analysis Plan Amendment 5 |
|---|---|
| Objectives | Endpoints |
| | The frequencies and percentages of participants with SAEs, AEs leading to withdrawal and AESIs throughout the study period: |
| | – Day 1 through Day 211 in cel |
| | – Day 1 through Day 241 in cel<br>groups, and |
| | – Day 1 through Day 361 in col |
| Phase II – Formulation | and Schedule-finding |
| | ndary |
| To describe the distribution of participants by percentages of serogroup B invasive disease strains killed using enchSBA at 1 month after the last vaccination of the vaccine (CCI) vaccine (CCI) administered at | The percentages of serogroup B invasive disease strains killed using enc-hSBA in each participant sample at 1 month after the last vaccination (Day 211, Month 7) in all |
| 0,2 and 0,6-months schedule and of the MenB vaccine administered at 0,6-months schedule. | |
| To assess the immune response to the column vaccine (ccl ) administered at 0,2 and 0,6-months schedule and to the MenB vaccine administered at 0.0 constitutions and the schedule and the schedul | The percentages of participants with hSBA titres ≥LLOQ for each and all serogroup B indicator strains at: |
| 0,6-months schedule against serogroup B indicator strains. | <ul> <li>Day 1, Month 0 in COL</li> <li>and Control groups,</li> </ul> |
| | - 3 months pre-first column vaccination (Day 31, Month 1) in column groups and, |
| | 1 month after the last vaccination (Day 211, Month 7) for all study groups. |
| | The percentages of participants with 4-fold rise in hSBA titres** at 1 month after the last vaccination for all study groups (Day 211, Month 7), relative to: |
| | Day 1, Month 0 for equations and, and Control groups and, |
| | - 3 months pre-first ccl vaccination (Day 31, Month 1) for ccl groups. |
| | hSBA GMTs against serogroup B indicator strains at: |
| | <ul> <li>Day 1, Month 0 in column and Control groups,</li> </ul> |
| | - 3 months pre-first column vaccination (Day 31, Month 1) in column groups and, |
| | 1 month after the last vaccination (Day 211, Month 7) for all study groups. |
| | <ul> <li>hSBA GMRs against serogroup B indicator strains at<br/>1 month after the last vaccination (Day 211, Month<br/>7) for all study groups relative to:</li> </ul> |

| Objectives | 1 | Statistical Analysis Plan Amendment t |
|---|---|---|
| Objectives | | Endpoints |
| | | <ul> <li>Day 1, Month 0 for oct</li> <li>and Control groups and</li> </ul> |
| | | - 3 months pre-first cci vaccination |
| | | (Day 31, Month 1) for CCI |
| | | groups. |
| To assess the immune response to the col | • | The percentages of participants with hSBA titres |
| vaccine (CCI) administered at 0,2 and 0,6- | | ≥LLOQ for serogroups A, C, W and Y at: |
| months schedule and to the MenACWY vaccine (single dose) against serogroups A, C, W and Y. | | <ul> <li>Day 1, Month 0 in CCI</li> </ul> |
| accept against corogroups 71, 6, 17 and 11. | | and Control groups, |
| | | - 3 months pre-first column vaccination |
| | | (Day 31, Month 1) in <b>CCI</b> groups, |
| | | <ul><li>1 month after the first ccl</li></ul> |
| | | vaccination (Day 31, Month 1) in the |
| | | ccl groups, |
| | | <ul> <li>1 month after the last col</li> </ul> |
| | | vaccination (Day 211, Month 7) for all ABCWY groups and, |
| | | <ul> <li>1 month after the MenACWY vaccination in</li> </ul> |
| | | the Control group (Day 31, Month 1). |
| | • | The percentages of participants with 4-fold rise in |
| | | hSBA titres** for serogroups A, C, W and Y at 1 |
| | | month after the first column vaccination (Day |
| | | 31, Month 1) relative to Day 1, Month 0 for groups. |
| | | hSBA GMTs against serogroups A, C, W and Y at: |
| | | • • • |
| | | <ul> <li>Day 1, Month 0 in ccl</li> <li>and Control group,</li> </ul> |
| | | - 3 months pre-first ccl vaccination |
| | | (Day 31, Month 1) in ccl |
| | | groups, |
| | | - 1 month after the first col |
| | | vaccination (Day 31, Month 1) in the groups, |
| | | <ul><li>1 month after the last CI</li></ul> |
| | | vaccination (Day 211, Month 7) for all ABCWY |
| | | groups and, |
| | | <ul> <li>1 month after the MenACWY vaccination in</li> </ul> |
| | | the Control group (Day 31, Month 1). |
| | • | hSBA GMRs against serogroups A, C, W and Y at 1 month after: |
| | | <ul> <li>the first ccl vaccination (Day 31,</li> </ul> |
| | | Month 1) in the CCI |
| | | groups, |
| | | <ul> <li>the last column vaccination (Day 211,<br/>Month 7) for all ABCWY groups and</li> </ul> |
| | | , |
| | | <ul> <li>the MenACWY vaccination in the Control<br/>group (Day 31, Month 1),</li> </ul> |
| | | group (Day O1, Month 1), |

| | Statistical Analysis Plan Amendme | |
|---|---|---|
| Objectives | Endpoints | |
| | relative to Day 1, Month 0 for column and Control groups and 3 months pre-first column vaccination (Day 31, Month 1) for column groups. The total IgG as measured by ELISA GMCs against serogroups A, C, W and Y at: | |
| | | <ul> <li>Day 1, Month 0 in column</li> <li>and Control groups,</li> </ul> |
| | | - 3 months pre- first class vaccination (Day 31, Month 1) in colamost |
| | | 1 month after the first column vaccination in the column groups and after the |
| | | MenACWY vaccination in the Control group (Day 31, Month 1) and, |
| CCI | | <ul> <li>1 month after the last CO vaccination (Day 211, Month 7) for all ABCWY groups.</li> </ul> |

212458 (MENACWY=colored -001 PRI) Statistical Analysis Plan Amendment 5



Abbreviations: AE, Adverse event; SAE, Serious adverse event; AESI, Adverse event of special interest; ELISA, enzyme-linked immunosorbent assay; GMC, geometric mean concentrations; enc-hSBA, endogenous complement human serum bactericidal assay; GMT, geometric mean titre; GMR, geometric mean ratio; hSBA, human serum bactericidal assay; LOD, limit of detection; LLOQ, lower limit of quantitation.

Note 1: MenB immune response will be assessed against N. meningitidis serogroup B indicator strains

Note 2: Evaluation of the tertiary objectives may or not be performed. If the tertiary objectives are evaluated, it may be assessed in a subset of participants using remaining serum after the primary and secondary analyses have been completed; no additional blood samples will be collected from participants.

<sup>\*</sup>All statistical criterion linked to evaluation of the objectives can be found in Section 9.4 in the protocol.

<sup>\*\*</sup>For the serogroup A C, W, Y and serogroup B evaluations, the 4-fold rise (for serogroup B - per each indicator strain) is defined in section 10.1.3.10.

<sup>&</sup>lt;sup>†</sup> The primary objective of immunological non-inferiority of the **CCI** vaccine to MenACWY will be evaluated only in participants without a previous MenACWY vaccination (unprimed). All other primary and secondary objectives will be evaluated in participants with and without previous MenACWY vaccination (primed and unprimed).

### 3. STUDY DESIGN

### 3.1. Overall design

This is a seamless Phase I/II multi-country, self-contained study comprising of 2 phases, in order to ensure the safety of participants.

### 3.1.1. Phase I study design

The Phase I safety lead-in will include 4 study groups (randomised 3:1), with a staggered enrolment (16 participants initially followed by 16 participants later) of a total of 32 participants (Figure 1).

- College : Participants will receive the College vaccine in a 0,1-month schedule.
- Participants will receive a saline placebo in a 0,1-month schedule, as control group for collection.
- Participants will receive the converge vaccine in a 0,1-month schedule.
- Participants will receive a saline placebo in a 0,1-month schedule, as control group for CO

For more detailed information on study groups and treatments administered, refer to Table 1.

Figure 1 Study design overview – Phase I (Safety Lead-in)



Abbreviation: N, number of participants; V, clinic visit; D, day; iSRC, internal safety review committee; PC, phone contact; BS, blood sample.

Note 1: This figure represents the main aspects of the study design. Refer to protocol Table 1 Schedule of activities, for details on all visits and contacts

Note 2: Refer to protocol Section 8 for information on study procedures during special circumstances.

29 Aug 2023 Page 17 of 48

212458 (MENACWY=ccl -001 PRI) Statistical Analysis Plan Amendment 5

Table 1 Study groups, intervention and blinding – Phase I

| Study groups | Number of participants | Age<br>(Min-Max) | Study intervention(s) | Blinding |
|---|---|---|---|---|
| CCI | 12 | 18-40 years | CCI | |
| | 12 | 18-40 years | | Observer blinded |
| | 4 | 18-40 years | NaCl | Observer-blinded |
| | 4 | 18-40 years | NaCl | |

**Duration of the Phase I of the study**: The intended duration of the Phase I of the study, per participant is approximately 7 months.

**Data collection**: Standardised Electronic Case Report Form (eCRF). Solicited events will be collected using a participant diary (electronic Diary [eDiary]).

#### Sampling schedule for Phase I of the study:

- Blood sample: An overall blood volume of *approximately* 240 mL per participant will be collected over the course of the Phase I part of the study, 80 mL at Visit 1 (Day 1), Visit 3 (Day 31) and Visit 4 (Day 61). An additional 7 mL of blood will be collected at Visit V1 and Visit V2 from all participants for the safety laboratory evaluation.
- Urine sample: Urine samples for pregnancy testing will be collected from female participants of childbearing potential at Visit 1 (Day 1) and Visit 3 (Day 31) prior to the study intervention.

### 3.1.2. Phase II study design

Phase II will start only after a positive outcome from the iSRC review of the safety data from participants receiving both vaccinations of the higher-dosage vaccine formulation in Phase I of the study. Phase II will be conducted in 2 parts: Formulation and Schedule-finding and Blood sourcing with enrolment commencing parallelly to both these parts.

#### 3.1.2.1. Phase II: Formulation and Schedule-finding

Phase II (Formulation and Schedule-finding) will include 5 study groups, with a staggered enrolment (45 participants for safety lead-in and 955 participants thereafter) of a total of 1000 participants (Figure 2):

- Participants will receive 2 vaccinations of the vaccine in a (0,6-months) schedule.
- Participants will receive 2 vaccinations of the vaccine in a (0,2-months) schedule.
- Participants will receive 2 vaccinations of the vaccine in a (0,6-months) schedule.
- Participants will receive 2 vaccinations of the vaccine in a (0,2-months) schedule.

212458 (MENACWY=ccl -001 PRI) Statistical Analysis Plan Amendment 5

The above 4 groups will also receive 1 injection of placebo, according to the schedule described in Figure 2.

• **Control**: Participants will receive 2 vaccinations of MenB vaccine (*Bexsero*) in a (0,6-months) schedule and a single vaccination of MenACWY vaccine (*Menveo*).

For more detailed information on study groups and treatments administered, refer to Table 2.

Figure 2 Study design overview – Phase II (Formulation and Schedule-finding)



Abbreviation: N, number of participants; V, clinic visit; D, day; TC, Telephone contact for Control group only; iSRC, internal safety review committee; PC, phone contact; BS, blood sample.

Note 1: Blood draw at Visit 6 Month 18 will be used only for assessment of tertiary objectives.

Note 2: This figure represents the main aspects of the study design.

Note 3: The Phase II (Formulation and Schedule-finding) is partially blinded. Study conduct and data collection in groups will be observer-blind while in group Control it will be open-label.

# # Day 121 Month 4 is a visit for CCI group (TC) When the second

Note 4: If local regulations allow and quality of study procedures is maintained, participant(s) can be offered remote visits (e.g., home visits) for the collection of biological samples and/or study intervention administration (except for Visit V1 which will always be a clinic visit). These remote visits must be performed by qualified study staff/ HCPs. Refer to the SoA (protocol Table 3) for the timing of these visits. Details of how these visits will be conducted are outlined in the SPM. Refer to protocol Section 8 (decentralised study procedures) for details

Note 5: Refer to protocol Section 8 for information on study procedures during special circumstances

<sup>^</sup> The phone call at Day 8 is only for the first 45 participants (15 participants in CCI and 5, 5 participants in CCI and 5 participants in the Control groups).

<sup>\*</sup> The outcome of the iSRC will impact the next study intervention at Month 4. The Month 1 blood sampling will proceed as planned

212458 (MENACWY=ccl -001 PRI)
Statistical Analysis Plan Amendment 5

A total of 45 participants will be randomised with 3:1:3:1:1 ratio to the 5 groups (15 in the CCI), 5 in the CCI), 5 in the CCI), 5 in the CCI), 5 in the CCI), 5 in the CCI), 5 in the CCI), 5 in the CCI), 6 in the CCI), 6 in the CCI), 7 in the CCI), 8 in the CC

Table 2 Study groups, intervention and blinding – Phase II (Formulation and Schedule-finding)

| Study groups | Number of participants | Age<br>(Min-Max) | Study intervention(s) | Blinding |
|---|---|---|---|---|
| CCI | 206 | 10 – 25 years | <mark>cci</mark><br>NaCl | |
| | 196 | 10 – 25 years | CCI<br>NaCl | Observer-blinded |
| | 206 | 10 – 25 years | CCI<br>NaCl | |
| | 196 | 10 – 25 years | CCI<br>NaCl | |
| Control | 196 | 10 – 25 years | MenACWY | Open label |
| | | | rMenB+OMV NZ | |

Duration of the Phase II (Formulation and Schedule-finding) of the study: The intended duration of the Phase II of the study, per participant is approximately 18 months.

**Data collection**: standardised eCRF. Solicited events will be collected using a participant diary (eDiary).

#### Sampling schedule for Phase II (Formulation and Schedule-finding) of the study:

• Blood sample: In order to provide the necessary serum volume for the bactericidal assays (enc-hSBA and/ or hSBA), an overall blood volume of *approximately* 90mL, per participant, will be collected over the course of the Phase II step of the study. Urine sample: Urine samples for pregnancy testing will be collected from female participants of childbearing potential at Visit 1 (Day 1), Visit 3 (Day 121) and Visit 4 (Day 181) prior to the vaccination in the ABCWY groups and at Visit 1 (Day 1) and Visit 4 (Day 181) prior to the vaccination in the Control group.

#### 3.1.2.2. Phase II: Sourcing

The blood sourcing part of the Phase II study will include 2 groups (randomised 1:1), with a parallel enrolment of a total of 226\* participants:

- Participants will receive 2 vaccinations of the vaccine in a (0,1-month) schedule.
- Participants will receive 2 vaccinations of the vaccine in a (0,1-month) schedule.

212458 (MENACWY=col -001 PRI) Statistical Analysis Plan Amendment 5

\* At the time of the protocol amendment to which this document refers (Protocol amendment 4), enrolment to these 2 groups had been stopped. The total number of participants enrolled have been presented in Figure 3.

Additionally, the Phase II sourcing part will include 4 more groups (randomised 1:1:1:1), with a parallel enrolment of a total of 240 participants (Figure 3):

- Participants will receive 2 vaccinations of the vaccine in a (0,2-month) schedule.
- Participants will receive 2 vaccinations of the vaccine in a (0,2-month) schedule.
- Participants will receive 2 vaccinations of the vaccine in a (0,6-month) schedule.
- Participants will receive 2 vaccinations of the vaccine in a (0,6-month) schedule.

For more detailed information on study groups and treatments administered, refer to Table 3.

The schedule of activities in the Phase II (sourcing) is described in Table 5, Table 6 and Table 7 in the protocol.

Figure 3 Study design overview – Phase II (Sourcing)

Abbreviation: N, number of participants; V, clinic visit; D, day, PC, phone contact; BS, blood sample.

Note 1: This figure represents the main aspects of the study design. Refer to protocol Table 5, Table 6 and Table 7, Schedule of activities, for details on all visits and contacts

Note 2: If local regulations allow and quality of study procedures is maintained, participant(s) can be offered remote visits (e.g., home visits) for the collection of biological samples and/or study intervention administration (except for Visit V1 which will always be a clinic visit). These remote visits must be performed by qualified study staff/ HCPs. Refer to

212458 (MENACWY=colored -001 PRI) Statistical Analysis Plan Amendment 5

the SoA (protocol Table 5, Table 6 and Table 7) for the timing of these visits. Details of how these visits will be conducted are outlined in the SPM. Refer to protocol Section 8 (decentralised study procedures) for details Note 3: Refer to protocol Section 8 for information on study procedures during special circumstances.

Table 3 Study groups, intervention and blinding – Phase II (Sourcing)

| Study groups | Number of participants | Age<br>(Min-Max) | Study intervention(s) | Blinding |
|---|---|---|---|---|
| - CCI | 107 | | CCI | |
| _ | 60<br>60 | 18-50 years | | Observer-<br>blinded* |
| _ | 60<br>60 | | | |

<sup>\*</sup> Due to the different vaccination schedules in Phase II Sourcing, the study will be observer blind only in terms of the vaccine formulations.

**Duration of the Phase II (Sourcing) of the study**: The intended duration of the Phase II (sourcing) of the study, per participant is:

- approximately 7 months for the column groups,
- approximately 8 months for the ccl groups, and,
- approximately 12 months for the column groups.

**Data collection**: Standardised Electronic Case Report Form (eCRF). Solicited events will be collected using a participant diary (electronic Diary [eDiary]).

### Sampling schedule for Phase II (Sourcing) of the study:

- Blood sample: An overall blood volume of *approximately* 285 mL per participant will be collected over the course of the Phase II, Sourcing part of the study. Urine sample: Urine samples for pregnancy testing will be collected from female participants of childbearing potential prior to the study intervention at the following timepoints:
  - at Visit 1 (Day 1) and Visit 2 (Day 31) for the groups,
  - at Visit 1 (Day 1) and Visit 2 (Day 61) for the groups, and,
  - at Visit 1 (Day 1) and Visit 2 (Day 181) for the groups.

The **primary completion date** for the study is the Day 541, Month 18 timepoint in Phase II. Refer to Protocol Section 9.4.6 for the planned interim analysis.

### 4. ANALYSIS SETS







212458 (MENACWY=ccl -001 PRI) Statistical Analysis Plan Amendment 5



### 5. STATISTICAL ANALYSES

Standard data derivation rules and stat methods are described in section 10.1 while the study specific data derivation rules and stat methods are described in section 9.

### 5.1. Disposition of subjects

### 5.1.1. Analysis of disposition of subjects

Number of subjects enrolled, vaccinated subjects (at least 1 vaccination, full vaccination course), reason for early withdrawal, FAS, and PPS will be described by vaccine group.

### 5.2. Analysis of demography and baseline characteristics

### 5.2.1. Analysis planned in the protocol

Demography and baseline characteristics analysis are not described in the protocol.

212458 (MENACWY=ccl -001 PRI) Statistical Analysis Plan Amendment 5

#### 5.2.2. Additional considerations

Descriptive statistics (mean, standard deviation, median, minimum and maximum) for age, height, weight, and body mass index (BMI) at enrolment will be calculated overall and by vaccine group.

Distributions of subjects by sex, race, ethnic origin will be summarised overall and by vaccine group.

### 5.3. Primary endpoints





212458 (MENACWY=cci -001 PRI)





### 5.3.2. Additional considerations

NA



- 5.4. Secondary endpoints
- 5.4.1. Analysis planned in the protocol
- 5.4.1.1. Phase I (Safety Lead-in)

NA

212458 (MENACWY=cci -001 PRI)



212458 (MENACWY=cci -001 PRI) Statistical Analysis Plan Amendment 5

## 5.4.1.3. Phase II (Sourcing)

NA
212458 (MENACWY=cci -001 PRI)



212458 (MENACWY=cci -001 PRI) Statistical Analysis Plan Amendment 5

212458 (MENACWY=cci -001 PRI) Statistical Analysis Plan Amendment 5

212458 (MENACWY=cci -001 PRI) Statistical Analysis Plan Amendment 5

212458 (MENACWY=set = -001 PRI)
Statistical Analysis Plan Amendment 5



# 9.1. Data derivation

NA

212458 (MENACWY=cci -001 PRI) Statistical Analysis Plan Amendment 5

9.2. Statistical method

NA

9.2.1. Adjusted GMT ratios

NA

9.2.2. Vaccine efficacy

NA

10. ANNEXES





#### 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

#### 10.1.2.3. Daily recording of solicited events

#### 10.1.2.3.1. Studies with electronic diaries

For studies using electronic diaries for the collection of solicited events, a solicited event will be considered present only when a daily recording of grade 1 or more is present.

#### 10.1.2.4. Unsolicited adverse events

Unsolicited adverse event summaries are including serious adverse events unless specified otherwise.

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' when displayed in a statistical output.

#### 10.1.3. Data derivation

#### 10.1.3.1. Age at first dose in days

When age at first dose is to be displayed in days, it will be calculated as:

Age = date of first dose minus date of birth

#### 10.1.3.2. Age at first dose in months

When age at first dose is to be displayed in months, it will be calculated as the number of complete calendar months between the date of birth (DOB) and the date of first dose. For example:

DOB = 
$$10JUN2017$$
, Date of first dose =  $10JUL2018 \rightarrow Age = 13$  months

### 10.1.3.3. Age at first dose in years

When age at first dose is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of first dose. For example:

#### 10.1.3.4. Weight

Weight will be presented in kilograms. Weights reported in pounds will be converted as follows:

Weight in kilograms = Weight in pounds / 2.2

#### 10.1.3.5. Height

Height will be presented in centimetres. Heights reported in feet and inches will be converted as follows:

Height in centimetres = Height in inches  $\times 2.54$ 

#### 10.1.3.6. Body mass index (BMI)

BMI will be calculated as follows:

BMI = (Weight in kilograms) / (Height in meters)
$$^2$$

## 10.1.3.7. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

# 10.1.3.8. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off | value |
| All other cases | missing |

#### 10.1.3.9. Geometric mean titres (GMTs) and concentrations (GMCs)

Geometric Mean Titre (GMT) or Concentration (GMC) calculations are performed by taking the inverse logarithm of the mean of the log titre or concentration transformations. Antibody titres or concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT/GMC calculation. Cut-off values are defined by the laboratory before the analysis.

#### 10.1.3.10. Calculation of the 4-fold rise

The 4-fold rise for serogroups A, C, W, Y and for serogroup B indicator strains is defined as:

- a post-vaccination hSBA titre ≥4 times the LOD or ≥LLOQ, whichever is greater, for subjects with a pre-vaccination hSBA titre <LOD,
- a post-vaccination hSBA titre ≥4 times the LLOQ for subjects with a pre-vaccination hSBA titre ≥LOD but <LLOQ, and
- a post-vaccination hSBA titre ≥4 times the pre-vaccination titre for subjects with a pre-vaccination hSBA titre ≥LLOQ.

The LOD and the LLOQ depend on the serogroup and the indicator strain, and are still under evaluation while this document is being amended.

#### 10.1.3.11. Onset day

The onset day for an event (e.g., AE, concomitant medication/vaccination) is the number of days between the last study dose and the start date of the event. This is 1 for an event occurring on the same day as a study dose (and reported as starting after study dose).

212458 (MENACWY=colored -001 PRI) Statistical Analysis Plan Amendment 5

#### 10.1.3.12. Duration of events

The duration of an event with a start and end date will be the difference between the start and end date plus one day, i.e., an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

# 10.1.3.13. Counting rules for combining solicited and unsolicited adverse events

Unsolicited adverse events with missing administration site flag will be considered systemic.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

#### 10.1.3.14. Counting rules for occurrences of solicited events

When the occurrences of solicited events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. In case of multiple reporting for the same solicited adverse event, the worst reported grade will be considered.

At visit 1 of Control group in Phase II F&SF two vaccines are injected, one in either arm. Therefore, administration site adverse events imputed during the first seven days after visit 1 must be related to a specific arm and vaccine. For subjects where, instead, it is not possible to uniquely associate one or more records of administration site adverse events to one of the two vaccines, then all the administration site events recorded by those subjects during the first seven days after vaccination will be excluded from the analysis. In this way, ambiguous records will not contribute to the denominator – nor to the numerator – when calculating frequencies and percentages of administration site adverse events at visit 1 of Control group. Systemic adverse events will still be reported as usual, as their records are never associated to a specific arm.

# 10.1.4. Display of decimals

### 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 subjects in each tabulated group
- one decimal when there are at least 50 subjects in at least one tabulated group
  - Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

212458 (MENACWY=colored -001 PRI) Statistical Analysis Plan Amendment 5

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

- The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.
- Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

# 10.1.4.2. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with one more decimal than the maximum number used to display the individual percentages, for example the difference between two percentages displayed with one decimal will be displayed with two decimals.

#### 10.1.4.3. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (height, weight, body mass index (BMI), pre-dose body temperature) will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maxima and minima of transformed height/weight variables will be displayed without decimals, with the exception of infant studies where one decimal will be displayed for the transformed weight.

The maximum and minimum of transformed body temperatures will be displayed with one decimal.

# 10.1.4.4. Serological summary statistics

The number of decimals used when displaying geometric mean titres (GMT) or concentrations (GMC) and their confidence limits is shown in the following table:

| GMT or GMC value | Number of decimals to display |
|------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT or GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e., the one with the higher number of decimals). For example, if GMT or GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

GMT or GMC group ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.



# 11. REFERENCES

